CLINICAL TRIAL: NCT01723072
Title: A Randomized, Double-blind, Placebo-controlled, 28-week Treatment With a 8 Week Follow-up to Investigate the Impact of Omalizumab on Quality of Life Measures and the Incidence and Severity of Angioedema Despite H1-antihistamine Therapy.
Brief Title: Impact of Omalizumab on Quality of Life Measures and Angioedema Occurrence in Patients With CSU Refractory to Therapy
Acronym: X-ACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIGE025EDE16
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Chronic Spontaneous Urticaria; Angioedema
Keywords: Chronic spontanous urticaria, refractory CSU, Angioedema
MeSH Terms: conditions — Chronic Urticaria; Angioedema | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Omalizumab (Experimental): omalizumab once a month via subcutaneous injection.
  Interventions: Biological: Omalizumab
- 2 Placebo (Placebo Comparator): placebo of omalizumab once a month via subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Omalizumab — Humanized monoclonal antibody against human IgE
  Other Names: IGE025
  Arms: 1 Omalizumab
Drug: Placebo — Placebo to omalizumab
  Other Names: Placebo for Omalizumab
  Arms: 2 Placebo

SUMMARY:
This study will assess the impact of omalizumab on the quality of life improvement when added to the standard therapy in refractory patients suffering from chronic spontaneous urticaria and angioedema.

DETAILED DESCRIPTION:
This study will be conducted using a double-blind, placebo-controlled, randomized, multicenter design to investigate the impact of omalizumab on Quality of Life (QoL) in Chronic Spontaneous Urticaria (CSU) and will assess its effectiveness in reducing and/or inhibiting the occurrence, time-course and severity of angioedema episodes.

Omalizumab is administered subcutaneously every 4 weeks as an add-on therapy to the current approved treatment of adult CSU patients. The treatment period is 28 weeks which is followed by an 8-week follow-up. The study aims to enroll approximately 70 patients.

The study is divided into a 2-week screening period, a 28-week double-blind treatment phase with omalizumab or placebo-omalizumab, and an 8-week follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic spontaneous urticaria (CSU) refractory to H1-antihistamine treatment
* Presence of itch an hives for more than 6 weeks
* UAS7 score of more than 14 (range 0-42)
* Patient has history of insufficient response to 4x of the approved dose of H1-antihistamines
* CSU diagnosis for more than 6 months
* Angioedema at least 4x in the last 6 months

Exclusion Criteria:

* Patients with non urticaria associated angioedema
* History of hypersensitivity to omalizumab or the rescue medication or to drugs of similar chemical structure
* Evidence of parasitic infection
* Previous treatment with omalizumab within the last 6 months prior to screening
* History of anaphylactic shock
* Woman who are pregnant or breast feeding
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-01-23 (Actual); Primary Completion 2014-05-09 (Actual); Study Completion 2014-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- Germany (24):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Selters
  - Novartis Investigative Site, Wiesbaden

REFERENCES:
- [Derived] Staubach P, Metz M, Chapman-Rothe N, Sieder C, Brautigam M, Canvin J, Maurer M. Effect of omalizumab on angioedema in H1 -antihistamine-resistant chronic spontaneous urticaria patients: results from X-ACT, a randomized controlled trial. Allergy. 2016 Aug;71(8):1135-44. doi: 10.1111/all.12870. Epub 2016 Mar 31. PMID 27010957

RESULTS

PARTICIPANT FLOW:
Groups:
- Omalizumab: Omalizumab once a month via subcutaneous injection.
- Placebo: Placebo of omalizumab once a month via subcutaneous injection
Period: Overall Study
Arm/Group | Omalizumab | Placebo
Started | 44 (28-week treatment period and 8-week follow-up period) | 47 (28-week treatment period and 8-week follow-up period)
Completed | 33 | 26
Not Completed | 11 | 21
Not completed — Withdrawal by Subject | 7 | 13
Not completed — Discon for rescue medication after wk 24 | 0 | 5
Not completed — Other | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 44 | 47 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (13.7) | 41.1 (10.6) | 42.9 (12.3)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 41 | 47 | 88
  >=65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 63
  Male | 14 | 14 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 42 | 46 | 88
  Asian | 1 | 1 | 2
  Other | 1 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 27.3 (6.3) | 29.0 (5.9) | 28.2 (6.1)
BMI group [Count of Participants; unit: Participants] — Body Mass Index group
  Participants
    <18.5 | 0 | 0 | 0
    18.5-25 | 20 | 12 | 32
    >25 | 24 | 35 | 59
Smoking status [Count of Participants; unit: Participants]
  Never smoked | 18 | 13 | 31
  Current smoker | 19 | 18 | 37
  Ex-smoker | 7 | 16 | 23
Disease history and baseline characteristics of angioedema (FAS) [Count of Participants; unit: Participants] — Frequency of prior angioedema episodes
  Participants
    Daily | 3 | 6 | 9
    Weekly | 21 | 24 | 45
    >6 episodes per year | 19 | 14 | 33
    <6 episodes a year | 1 | 3 | 4
[Disease history and baseline characteristics of angioedema (FAS)] [Count of Participants; unit: Participants] — Duration of symptoms of angioedema (usually)
  Participants
    <24 hours | 25 | 25 | 50
    >24 hours | 19 | 22 | 41
Disease history and baseline characteristics of angioedema (FAS) [Number; unit: participants] — Location of prior angioedema (any)
  participants
    Eyes/lids/periorbital | 36 | 41 | 77
    Lips/perioral | 37 | 41 | 78
    Mouth/laryngeal | 22 | 28 | 50
    Trunk | 10 | 20 | 30
    Arms/legs | 24 | 28 | 52
    Hands | 27 | 34 | 61
Disease history and baseline charactaristics [Mean (Standard Deviation); unit: years] — Duration of disease before baseline
  years | 8.4 (9.3) | 7.4 (8.8) | 7.9 (9.0)
Disease history and baseline charactaristics [Count of Participants; unit: Participants] — Duration of disease group - n
  Participants
    <2 years | 13 | 13 | 26
    2-10 years | 18 | 27 | 45
    >10 years | 13 | 7 | 20
Disease history and baseline charactaristics [Count of Participants; unit: Participants] — Previous systemic corticosteroid use - n
  Participants
    No | 33 | 32 | 65
    Yes | 11 | 15 | 26
Disease history and baseline charactaristics [Count of Participants; unit: Participants] — Previous number of nsH1-n antihistamines - n
  Participants
    <=2 years | 42 | 40 | 82
    3-5 years | 2 | 7 | 9
    >5 years | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline Using Chronic Urticaria Quality of Life Questionnaire (CU-Q2oL) Total Scores During the Study: Unadjusted Analysis and ANCOVA (LOCF) (FAS)
Description: The CU-Q2oL is a questionnaire that measures the relative burden of chronic urticaria on subjective well-being. It consists of 23 questions in 3 domains (symptoms, general impairment, difficulties and problems due to urticaria). Participants are asked to respond how much they are troubled by each problem on a 5-point Likert scale (1= not at all to 5= very much). An overall score is calculated and normalized to a scale of 1 to 100.
Time Frame: Baseline, 4, 12, 20, 28 and 36 weeks
Population: full analysis set
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 44 | 47
score
  V3 (week 4) | -25.5 (21.3) | -6.4 (15.9)
  V5 (week 12) | -32.1 (21.8) | -12.1 (20.3)
  V7 (week 20) | -31.4 (23.7) | -16.2 (18.8)
  V9 (week 28) | -35.1 (24.2) | -13.9 (17.7)
  Follow-up (week 36) | -23.9 (23.0) | -14.7 (19.2)

2. Secondary Outcome: Number of Angioedema Burdened Days by Study Phase (Observed Cases With Imputation)
Time Frame: Baseline, week 28; and the follow-up period (weeks 29-36)
Population: full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 44 | 47
days
  Screening (Week -2 to -1) | 5.2 (3.9) | 6.8 (4.3)
  Treatment (Week 1 to 28) | 14.6 (19.5) | 49.5 (50.8)
  Follow-up (Week 29 to 36) | 5.8 (9.1) | 12.8 (16.2)

3. Secondary Outcome: Mean Time Interval Between Successive Angioedema Episodes of the First 15 Episodes
Time Frame: Baseline to week 28
Population: full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 44 | 47
days
  1st to 2nd episode: number analyzed (Participants) | 36 | 43
  1st to 2nd episode | 20 (41.63) | 7.8 (14.29)
  2nd to 3rd episode: number analyzed (Participants) | 30 | 42
  2nd to 3rd episode | 11.0 (19.52) | 7.2 (10.16)
  3rd to 4th episode: number analyzed (Participants) | 28 | 39
  3rd to 4th episode | 26.4 (50.73) | 8.3 (13.24)
  4th to 5th episode: number analyzed (Participants) | 27 | 36
  4th to 5th episode | 14.9 (23.87) | 8.6 (20.44)
  5th to 6th episode: number analyzed (Participants) | 25 | 34
  5th to 6th episode | 14.2 (20.54) | 13.6 (30.09)
  6th to 7th episode: number analyzed (Participants) | 21 | 31
  6th to 7th episode | 11.2 (22.11) | 7.5 (11.32)
  7th to 8th episode: number analyzed (Participants) | 15 | 29
  7th to 8th episode | 18.1 (29.41) | 9.1 (17.58)
  8th to 9th episode: number analyzed (Participants) | 14 | 28
  8th to 9th episode | 10.7 (15.05) | 8.0 (12.26)
  9th to 10th episode: number analyzed (Participants) | 11 | 26
  9th to 10th episode | 11.4 (20.16) | 8.7 (12.26)
  10th to 11th episode: number analyzed (Participants) | 11 | 23
  10th to 11th episode | 11.5 (13.02) | 8.5 (10.41)
  11th to 12th episode: number analyzed (Participants) | 10 | 21
  11th to 12th episode | 8.9 (9.42) | 9.4 (13.89)
  12th to 13th episode: number analyzed (Participants) | 8 | 18
  12th to 13th episode | 6.0 (4.47) | 4.3 (4.43)
  13th to 14th episode: number analyzed (Participants) | 8 | 18
  13th to 14th episode | 3.6 (3.02) | 7.3 (4.56)
  14th to 15th episode: number analyzed (Participants) | 7 | 17
  14th to 15th episode | 6.9 (9.96) | 10.1 (11.86)

4. Secondary Outcome: Change of Angioedema Activity Score (AAS) Total Week Sum Scores: Unadjusted Analysis and ANCOVA (Observed Cases With Imputation)
Description: A cumulative activity score, evaluated in the screening period and throughout the study. The records each evening on a daily basis symptoms of itch and hives into a patient diary. min. score = 0 ; max. score= 100
Time Frame: Baseline to week 28; and follow-up period (to week 36)
Population: full analysis set
Measure: Mean (Standard Deviation); unit: AAS (Angioedema Activity Score)
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 44 | 47
AAS (Angioedema Activity Score)
  Diary week 4: number analyzed (Participants) | 43 | 44
  Diary week 4 | -17.7 (20.0) | -5.0 (18.2)
  Diary week 12: number analyzed (Participants) | 39 | 34
  Diary week 12 | -19.0 (22.4) | -9.0 (22.8)
  Diary week 20: number analyzed (Participants) | 35 | 32
  Diary week 20 | -21.3 (21.6) | -16.9 (21.0)
  Diary week 28: number analyzed (Participants) | 34 | 32
  Diary week 28 | -20.6 (21.5) | -10.8 (21.3)
  Diary week 36: number analyzed (Participants) | 23 | 16
  Diary week 36 | -9.6 (18.4) | -15.3 (20.8)

5. Secondary Outcome: Diameter: Acute Swelling Episodes Within the Screening Period (Week -2 to -1)
Description: data points per group
Time Frame: week -2 to -1
Population: full analysis set
Measure: Number; unit: Number of episodes
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 44 | 47
Number of episodes
  Acute swelling episode, Diameter <10cm | 146 | 165
  Acute swelling episode, Diameter 10-20cm | 54 | 99
  Acute swelling episode, Diameter >20cm | 19 | 46
  unknown | 12 | 15

6. Secondary Outcome: Diameter: Acute Swelling Episodes at End of Treatment (Weeks 25 to 28)
Description: data points per group
Time Frame: weeks 25 to 28
Population: actual patient numbers
Measure: Number; unit: Number of episodes
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 34 | 25
Number of episodes
  Acute swelling episode, Diameter <10cm | 31 | 76
  Acute swelling episode, Diameter 10-20cm | 0 | 94
  Acute swelling episode, Diameter 20cm | 0 | 24
  unknown | 0 | 12

7. Secondary Outcome: Diameter: Acute Swelling Episodes at End of Follow-up(Weeks 33 to 36)
Description: data points per group
Time Frame: weeks 33 to 36
Population: full analysis set
Measure: Number; unit: Number of episodes
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 33 | 23
Number of episodes
  Acute swelling episode, Diameter <10cm | 92 | 90
  Acute swelling episode, Diameter 10-20cm | 28 | 58
  Acute swelling episode, Diameter >20cm | 8 | 19
  unknown | 17 | 18

8. Secondary Outcome: Shortness of Breath: Acute Swelling Episodes Within the Screening Period (Weeks -2 to -1)
Description: data points per group
Time Frame: weeks -2 to -1
Population: full analysis set
Measure: Number; unit: number of episodes
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 44 | 47
number of episodes
  Shortness of breath: No | 203 | 264
  Shortness of breath: Slightly | 13 | 25
  Shortness of breath: Moderately | 7 | 25
  Shortness of breath: Severely | 1 | 7
  Unknown | 7 | 4

9. Secondary Outcome: Shortness of Breath: Acute Swelling Episodes at End of Treatment Period (Weeks 25 to 28)
Description: data points per group
Time Frame: weeks 25 to 28
Population: full analysis set
Measure: Number; unit: Number of episodes
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 31 | 25
Number of episodes
  Shortness of breath: No | 28 | 195
  Shortness of breath: Slightly | 3 | 5
  Shortness of breath: Moderately | 0 | 5
  Shortness of breath: Severely | 0 | 0
  Unknown | 0 | 1

10. Secondary Outcome: Shortness of Breath: Acute Swelling Episodes at End of Follow-up Period (Weeks 33 to 36)
Description: data points per group
Time Frame: weeks 33 to 36
Population: full analysis set
Measure: Number; unit: Number of episodes
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 145 | 185
Number of episodes
  Shortness of breath: No | 127 | 172
  Shortness of breath: Slightly | 14 | 5
  Shortness of breath: Moderately | 1 | 3
  Shortness of breath: Severely | 0 | 1
  Unknown | 3 | 4

11. Secondary Outcome: Change of AE-Q2oL Scores From Baseline to Week 28: Unadjusted Analysis and ANCOVA (Observed Cases)
Description: The AE-Q2oL is a questionnaire for patients suffering from angioedema. It consists of 29 questions relevant to angioedema and its specific impact on quality of life. Patients are asked to respond how much they are troubled be each problem on a 5-point Likert scale (1= does not apply to 5= very much). An overall score is calculated and a higher score indicates lower quality of life. A negative change score (week 28 score minus baseline score) indicates improvement.
  Each AE-QoL question has 5 answer options (scored 1-5), with lower and higher scores indicting less and more adverse impact, respectively. The total score is calculated, which is then transformed into a linear scale that ranges from 0 to 100, with a score of 100 indicating the worst possible impairment of HRQoL
Time Frame: baseline to week 28; and then follow-up to week 36
Population: full analysis set
Measure: Mean (Standard Deviation); unit: AE-QoL Score
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 44 | 47
AE-QoL Score
  week 4 (n=38,36): number analyzed (Participants) | 38 | 36
  week 4 (n=38,36) | -26.5 (20.4) | -10.3 (21.0)
  week 12 (n= 35, 29): number analyzed (Participants) | 35 | 29
  week 12 (n= 35, 29) | -37.4 (23.8) | -20.4 (27.4)
  week 20 (n=34,27): number analyzed (Participants) | 34 | 27
  week 20 (n=34,27) | -37.1 (26.5) | -28.8 (22)
  week 28 (n=34, 25): number analyzed (Participants) | 34 | 25
  week 28 (n=34, 25) | -41.4 (25.7) | -24.2 (24.3)
  follow-up, week 36 (n=33,23): number analyzed (Participants) | 33 | 23
  follow-up, week 36 (n=33,23) | -27.2 (26.4) | -24.6 (23.3)

12. Secondary Outcome: Rescue Medication During the Treatment Period
Time Frame: baseline to 28 weeks
Population: safety set
Measure: Number; unit: participants
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 44 | 47
participants
  Any rescue medication | 25 | 35
  Any nsH1 - antihistamine rescue medication | 19 | 27
  Any clemastine rescue medication | 12 | 26
  Any corticosteroid rescue medication | 5 | 13
  Betamethasone | 2 | 12
  Prednisolone | 3 | 3
  Prednisolone succinate | 2 | 0

13. Secondary Outcome: Days of Rescue Medication During the Treatment Period
Description: data points per group
Time Frame: baseline to 28 weeks
Population: safety set
Measure: Number; unit: days
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 44 | 47
days
  Any rescue medication | 507 | 787
  Any nsH1 - antihistamine rescue medication | 403 | 524
  Any clemastine rescue medication | 92 | 236
  Any corticosteroid rescue medication | 25 | 113

14. Secondary Outcome: Days of Rescue Medication During the Follow-up Period
Description: data points per group
Time Frame: weeks 33 to 36
Population: safety set
Measure: Number; unit: days
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 44 | 47
days
  Any rescue medication | 165 | 118
  Any nsH1 - antihistamine rescue medication | 158 | 85
  Any clemastine rescue medication | 15 | 19
  Any corticosteroid rescue medication | 0 | 17

15. Secondary Outcome: Change of UAS7 Total Scores From Baseline to Week 28: Unadjusted Analysis and ANCOVA (Observed Cases)
Description: The UAS7 is the sum of urticaria activity scores over a seven day period. The possible range of the weekly UAS7 score is 0-42. 0 means complete response and a better outcome and 42 means no response and a worse outcome.
  Complete UAS7 response is defined as UAS7=0. The UAS7 is the sum of the Hive Severity Score over seven days (HSS7) and the Itch Severity Score over seven days (ISS7) . The Hive Severity Score has a scale of 0 (none) to 3 (intense/severe). Complete hives response is defined as HSS7=0. The Itch Severity Score has a scale of 0 (None) to 3 (Severe (difficult to tolerate)). Complete itch response is defined as ISS7=0
Time Frame: baseline to week 28; and then follow-up to week 36
Population: full analysis set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 44 | 47
scores on a scale
  week 4 | -12.6 (13.3) | -3.0 (9.4)
  week 12 | -16.4 (14.3) | -4.4 (13.3)
  week 20 | -15.0 (15.0) | -7.2 (14.7)
  week 28 | -16.8 (14.8) | -6.5 (13.4)
  follow-up, week 36 | -8.3 (15.3) | -6.2 (13.3)

16. Secondary Outcome: Change of DLQI Scores From Baseline to Week 28: Unadjusted Analysis and ANCOVA (Observed Cases)
Description: change in Dermatology Quality of Life Index scores
  The DLQI is a ten item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases such as eczema, psoriasis, acne and viral worts. It is a self-administered questionnaire which includes domains of daily activity, leisure, personal relationships, symptoms and feelings, treatment and school/work activities. Each domain has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is a valid score also and is scored as 0. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment.
Time Frame: baseline to week 28; and follow-up to week 36
Population: full analysis set
Measure: Mean (Standard Deviation); unit: DLQI Score
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 44 | 46
DLQI Score
  week 4 | -8.3 (7.3) | -2.4 (6.9)
  week 12 | -10.1 (7.5) | -3.9 (7.6)
  week 20 | -9.5 (8.4) | -5.1 (8.3)
  week 28 | -10.5 (8.3) | -5.6 (8.0)
  follow-up, week 36 | -6.8 (8.6) | -5.4 (8.3)

ADVERSE EVENTS:
Arm/Group | Omalizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 4/44 | 2/47
Other Adverse Events (participants affected / at risk) | 19/44 | 29/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=44) | Placebo (N=47)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=44) | Placebo (N=47)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 2 | 2
Pyrexia (General disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 9 | 13
Sinusitis (Infections and infestations) | 2 | 0
Hepatic enzyme increased (Investigations) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 4 | 4
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 6
Hypertension (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Publications from a single-site are postponed until publication of the pooled clinical trial data (i.e., data from all sites) or disclosure of trial results in their entirety.